CLINICAL TRIAL: NCT06956404
Title: Transcranial Photobiomodulation in Older Adults With Traumatic Brain Injury: Effects on Cerebral Blood Flow and Cognition
Brief Title: tPBM in Older Adults With Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-00956; CDMRP-TP230318 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury
Keywords: TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tPBM (Experimental): Subjects complete 18 t-PBM treatments, ~12 min per day, 3 days per week, for 6 weeks. tPBM will be administered via continuous, 808 nm wavelength laser delivery to the forehead at the standard scalp location.
  Interventions: Device: Transcranial photobiomodulator (tPBM)
- Sham tPBM (Sham Comparator): Subjects complete 18 sham treatments, ~12 min per day, 3 days per week, for 6 weeks. The sham treatment will be administered to the forehead at the standard scalp location.
  Interventions: Device: Transcranial photobiomodulator (tPBM) in sham mode

INTERVENTIONS:
Device: Transcranial photobiomodulator (tPBM) — The tPBM-2.0 device consists of a therapeutic laser console (that produces laser energy as NIR), and an optical delivery system consisting of a flexible, double-sheathed optical fiber connected to a custom helmet (cap). tPBM will be administered via continuous, 808 nm wavelength laser delivery to the forehead at the standard scalp location ~12 minutes per day, 3 days per week, for 6 weeks (18 total sessions).
  Other Names: Transcranial PhotoBioModulation-1000 (tPBM-2.0)
  Arms: Active tPBM
Device: Transcranial photobiomodulator (tPBM) in sham mode — The tPBM-2.0 device consists of a therapeutic laser console (which will be in sham mode, which does not produce laser energy), and an optical delivery system consisting of a flexible, double-sheathed optical fiber connected to a custom helmet (cap).
  Other Names: Transcranial PhotoBioModulation-1000 (tPBM-2.0)
  Arms: Sham tPBM

SUMMARY:
The purpose of this study is to evaluate the effect of transcranial photobiomodulation (tPBM) in older patients with chronic traumatic brain injury (TBI). The study aims to examine the effect of tPBM on prefrontal cerebral blood flow (CBF) and executive function (EF)

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent and follow study procedures.
2. Age ≥ 55 years and ≤ 85 years.
3. History of non-penetrating TBI of at least moderate severity,

   1. defined by Emergency Department Glasgow Coma Scale (GCS) < 13,
   2. or post-traumatic amnesia > 24 hours,
   3. or loss of consciousness > 30 minutes,
   4. or evidence of trauma-related abnormality on acute neuroimaging.
4. Between 1 and 2 years post injury.

Exclusion Criteria:

1. Delayed loss of consciousness due to expanding lesions
2. Diagnosis of dementia, history of brain tumor, or other serious neurological disorder
3. Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnosis of alcohol or drug use disorder or history of other major psychiatric illness diagnosed with Mini-International Neuropsychiatric Interview (MINI)
4. History of significant cardiovascular or cerebrovascular pathology before sustaining TBI
5. Unstable medical conditions or medications impacting cognition (e.g., topiramate)
6. Significant skin conditions on the subject's scalp in the area of illumination
7. Large bilateral prefrontal cortex (PFC) lesions (i.e., more than 50% of our middle frontal gyrus region of interest (ROI) in both hemispheres)
8. Claustrophobia or metallic foreign bodies that would preclude MRI
9. Unwilling/unable to comply with study as judged by the Principal Investigator
10. Body mass index > 40 kg/m2 to fit comfortably in MRI
11. Past intolerance or hypersensitivity to tPBM
12. Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in prefrontal Cerebral Blood Flow (CBF) | Baseline, end-of-treatment (up to 6 weeks)
  CBF will be demonstrated by using arterial spin-labeled (ASL) magnetic resonance imaging (MRI), a method that can reliably quantify absolute CBF level across longer time intervals
Change in Executive Function (EF) composite scores | Baseline, end-of-treatment (up to 6 weeks)
  EF composite scores will be derived from five neuropsychological tests (Repeatable Battery for the Assessment of Neuropsychological Status - RBANS, Stroop Color-Word Test, Controlled Oral Word Association Test/FAS, Trail Making Test-A& B) that assess various aspects of EF.

SECONDARY OUTCOMES:
Change in number of treatment emergent adverse events as measured by the Systematic Assessment for Treatment Emergent Effects-Systematic Inquiry (SAFTEE-SI) | Baseline, end-of-treatment (up to 6 weeks)
  The SAFTEE-SI is a commonly used instrument originally developed by National Institute of Mental Health (NIMH) and adapted into a self-report instrument. The scale examines in a systematic fashion all possible treatment-emergent side effects and probes specific adverse symptoms, including suicidal thoughts and behaviors, and self-injurious behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Bushnik, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: jkim@med.cuny.edu. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to jkim@med.cuny.edu. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.